CLINICAL TRIAL: NCT06560996
Title: Effects of Short-term Very Low-calorie Diets on Cardiometabolic Health Markers in Humans
Brief Title: Very Low-calorie Diet & Cardiometabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Chenot Group, HC International SA (Unknown)
Responsible Party: Principal Investigator, Kostas Tsintzas, Professor of Human Physiology, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: FMHS 67-1123
Record Dates: First submitted 2024-06-26; First posted 2024-08-19 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Fasting; Cardiometabolic health; Autophagy
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): 7 days isoenergetic (weight maintaining) diet
- Very low calorie diet with low protein content (VLCD-LP group) (Experimental): 7 days very low-calorie diet (850 kcal per day) with low protein content (10% energy from protein, 45% from carbohydrate and 45% from plant-based fat)
  Interventions: Other: Very low calorie diet with low protein content (VLCD-LP group)
- Very low calorie diet with high protein content (VLCD-HP group) (Experimental): 7 days very low-calorie diet with high protein content (30% energy from protein, 45% from carbohydrate and 25% from plant-based fat)
  Interventions: Other: Very low calorie diet with high protein content (VLCD-HP group)

INTERVENTIONS:
Other: Very low calorie diet with low protein content (VLCD-LP group) — Very low calorie diet (850 kcals per day) with low protein content (10%)
  Arms: Very low calorie diet with low protein content (VLCD-LP group)
Other: Very low calorie diet with high protein content (VLCD-HP group) — Very low calorie diet (850 kcals per day) with high protein content (30%)
  Arms: Very low calorie diet with high protein content (VLCD-HP group)

SUMMARY:
To investigate the effects of a short-term (1-week) nutritional intervention in healthy individuals using very low-calorie (fasting-mimicking) diets with different protein content on markers of cardiometabolic health and autophagy.

DETAILED DESCRIPTION:
The aim of this project is to investigate the metabolic effects of a short-term (1-week) nutritional intervention in healthy humans using very low-calorie (fasting-mimicking) diets with low and high protein content on key cardiometabolic outcomes (with blood glucose as a primary outcome) and autophagy, oxidative stress, inflammation, functional measures of cardiovascular health, body composition, and faecal markers for gut microbiome diversity (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Participant is willing and able to comply with the requirements of the study protocol
* Aged between 18 and 65 years
* Healthy individual

Exclusion Criteria:

* A BMI <18 or >35 kg/m2
* Regularly skipping breakfast
* On an energy-restricted diet
* Taking medication to control appetite
* Eating Attitudes Test (EAT-26) score >20 as self-reported marker of symptoms and concerns characteristic of eating disorders
* Active metabolic (e.g. diabetes), endocrine (e.g. hyperthyroidism) or cardiovascular (e.g. heart or blood) abnormalities including hypertension or heart failure
* Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Fasting blood glucose | Day 0, Day 8
  To determine the impact of very low-calorie diets on fasting blood glucose concentration and the addition of low and high protein

SECONDARY OUTCOMES:
Measure circulatory autophagy marker Beclin-1 | Day 0, Day 8
  To determine the impact of very low-calorie diets with low and high protein content on Beclin-1 measured using Western Blotting and real-time polymerase chain reaction (PCR) techniques.
Measure circulatory autophagy marker Microtubule-associated protein 1A/1B-light chain 3 (LC3) | Day 0, Day 8
  To determine the impact of very low-calorie diets with low and high protein content on LC3 measured using Western Blotting and PCR techniques.
Measure circulatory autophagy proteins (ATGs) | Day 0, Day 8
  To determine the impact of very low-calorie diets with low and high protein content on ATGs measured using Western Blotting and real-time PCR techniques.
Measure cardiometabolic health via insulin levels | Day 0, Day 8
  To determine the impact of very low-calorie diets with low and high protein content on insulin using enzyme linked immunosorbant assays.
Measure circulatory inflammation via Insulin like-growth factor-1 (IGF-1) levels | Day 0, Day 8
  To determine the impact of very low-calorie diets with low and high protein content on serum IGF-1 levels using enzyme linked immunosorbant assays.
Measure circulatory inflammation via C-reactive protein levels | Day 0, Day 8
  To determine the impact of very low-calorie diets with low and high protein content on serum C-reactive protein levels using enzyme linked immunosorbant assays.
Measure circulatory inflammation via Tumour Necrosis factor alpha-1 (TNF-alpha) levels | Day 0, Day 8
  To determine the impact of very low-calorie diets with low and high protein content on serum TNFalpha levels using enzyme linked immunosorbant assays.
Measure of cardiovascular health with blood pressure | Day 0, Day 8
  To determine the impact of very low-calorie diets with low and high protein content on supine and standing blood pressure (both diastolic and systolic).
Functional measures of cardiovascular health | Day 0, Day 8
  To determine the impact of very low-calorie diets with low and high protein content on arterial stiffness using suprasternal notch-femoral pulse wave velocity by ArterioGraph.
Functional measures of cardiovascular health with heart rate | Day 0, Day 8
  To determine the impact of very low-calorie diets with low and high protein content on heart rate and heart rate variability.
Measures of cardiovascular health with autonomic function (blood pressure) | Day 0, Day 8
  To determine the impact of very low-calorie diets with low and high protein content on autonomic function (blood pressure [diastolic and systolic] response to postural change and rhythmic breathing).
Measures of cardiovascular health with autonomic function (heart rate) | Day 0, Day 8
  To determine the impact of very low-calorie diets with low and high protein content on autonomic function (heart rate response to postural change and rhythmic breathing).
Body composition | Day 0, Day 8
  To determine the impact of very low-calorie diets with low and high protein content on body fat mass and lean mass using DEXA (dual energy x-ray absorptiometry).
Faecal markers for gut microbiome diversity | Day 0, Day 8
  To determine the impact of very low-calorie diets with low and high protein content on microbiome diversity using stool analysis techniques (16S Metagenomic Sequencing)
Urine markers of protein metabolism | Day 0, Day 8
  To determine the impact of very low-calorie diets with low and high protein content on urinary markers of protein metabolism (ratio of urea to creatinine) using established biochemical (spectrophotometric) methods

CONTACTS AND LOCATIONS:
Overall Officials: Kostas Tsintzas, PhD, Principal Investigator — University of Nottingham
Locations (1):
- HC International SA, Weggis, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilhelmsen A, Davies A, Mallinson J, Pabla P, Jones R, Palmer EA, Dunn WB, Moran GW, Stephens FB, Tsintzas K. Acute effects of prior dietary fat ingestion on postprandial metabolic responses to protein and carbohydrate co-ingestion in overweight and obese men: A randomised crossover trial. Clin Nutr. 2022 Aug;41(8):1623-1635. doi: 10.1016/j.clnu.2022.06.022. Epub 2022 Jun 16. PMID 35764009
- [Background] Gao Y, Tsintzas K, Macdonald IA, Cordon SM, Taylor MA. Effects of intermittent (5:2) or continuous energy restriction on basal and postprandial metabolism: a randomised study in normal-weight, young participants. Eur J Clin Nutr. 2022 Jan;76(1):65-73. doi: 10.1038/s41430-021-00909-2. Epub 2021 May 26. PMID 34040199
- [Background] Jones R, Pabla P, Mallinson J, Nixon A, Taylor T, Bennett A, Tsintzas K. Two weeks of early time-restricted feeding (eTRF) improves skeletal muscle insulin and anabolic sensitivity in healthy men. Am J Clin Nutr. 2020 Oct 1;112(4):1015-1028. doi: 10.1093/ajcn/nqaa192. PMID 32729615
- [Background] Templeman I, Smith HA, Chowdhury E, Chen YC, Carroll H, Johnson-Bonson D, Hengist A, Smith R, Creighton J, Clayton D, Varley I, Karagounis LG, Wilhelmsen A, Tsintzas K, Reeves S, Walhin JP, Gonzalez JT, Thompson D, Betts JA. A randomized controlled trial to isolate the effects of fasting and energy restriction on weight loss and metabolic health in lean adults. Sci Transl Med. 2021 Jun 16;13(598):eabd8034. doi: 10.1126/scitranslmed.abd8034. PMID 34135111
- [Background] Gonzalez JT, Richardson JD, Chowdhury EA, Koumanov F, Holman GD, Cooper S, Thompson D, Tsintzas K, Betts JA. Molecular adaptations of adipose tissue to 6 weeks of morning fasting vs. daily breakfast consumption in lean and obese adults. J Physiol. 2018 Feb 15;596(4):609-622. doi: 10.1113/JP275113. Epub 2017 Dec 20. PMID 29193093
- [Derived] Burns L, Cooper S, Sarmad S, Funke G, Di Mauro A, Gaitanos GC, Tsintzas K. Effects of fasting-mimicking diets with low and high protein content on cardiometabolic health and autophagy: A randomized, parallel group study. Clin Nutr. 2025 Sep;52:299-312. doi: 10.1016/j.clnu.2025.08.004. Epub 2025 Aug 6. PMID 40816210